CLINICAL TRIAL: NCT05868057
Title: Clinical Studies Evaluating the Relative Bioavailability of SHR7280 Dry Suspension and Tablets (Single-center, Randomized, Open-label, Crossover)
Brief Title: A Clinical Study Evaluating the Relative Bioavailability of SHR7280 Dry Suspension and Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SHR7280-105
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis, Uterine Fibroids, Male Hormone-sensitive Prostate Cancer, Assisted Reproduction
MeSH Terms: conditions — Endometriosis; Leiomyoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group ARM 1 (Experimental): SHR7280 dry suspension then SHR7280 tablets
  Interventions: Drug: SHR7280 tablets; Drug: SHR7280 dry suspension
- Treatment group ARM 2 (Experimental): SHR7280 tablets, then SHR7280 dry suspension
  Interventions: Drug: SHR7280 tablets; Drug: SHR7280 dry suspension

INTERVENTIONS:
Drug: SHR7280 tablets — SHR7280 tablets 1 time
Drug: SHR7280 dry suspension — SHR7280 dry suspension 1 time

SUMMARY:
To assess the relative bioavailability of SHR7280 dry suspension and tablets in healthy subjects.

To assess the safety and tolerability of a single dose of SHR7280 dry suspension and tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before the start of the activities related to the trial, and be able to understand the procedures and methods of the trial, and be willing to strictly abide by the clinical trial protocol to complete the trial;
2. Age 18~45 years old (including both end values, subject to the signing of informed consent);
3. Male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI): 18~30 kg/m2 (including both end values);
4. Those who have no birth plan and no sperm or egg donation plan within 1 week after signing the informed consent form and the last dose, and agree to use highly effective contraceptive measures;
5. Women have regular menstruation in the last 3 days before the screening visit, with a menstrual cycle of 24~35 days and a menstrual period of 3~7 days.

Exclusion Criteria:

1. Female screening period or baseline period (D-1) urine pregnancy test or serum pregnancy test (serum β-HCG test) results are positive;
2. The female had any form of pregnancy (including spontaneous abortion, childbirth, ectopic pregnancy, etc.) within 3 months before randomization, or was breastfeeding at the time of the screening visit;
3. Women found ovarian cysts or masses with a diameter of ≥ 4 cm during the screening period;
4. Women use the following contraceptive methods during screening visits: drug sustained-release IUD, sustained-release contraceptives (subcutaneous implants, vaginal rings, microspheres and microcapsule contraceptive injections); Use of long-acting contraceptive injections before screening (contraindicated 3 months before screening for medroxyprogesterone acetate and 1 month before screening for other injections), oral contraceptives 2 months before screening, and contraceptives 1 month before screening; Special circumstances are judged by the investigator;
5. Those with a history of tobacco addiction in the previous 3 months (an average daily smoking > 5);
6. Average daily alcohol intake of more than 25 g (e.g., 750 mL of beer, 250 mL of wine, or 50 mL of liquor) in the 3 months prior to randomization;
7. Consumed any drink or food containing grapefruit within 7 days prior to randomization; or eat any beverage or food containing methylxanthines, such as coffee, tea, cola, chocolate, etc., within 2 days before randomization;
8. Allergic constitution, or suspected allergy to any ingredient in SHR7280 preparation;
9. Drug abusers, or positive urine drug abuse screening at screening, including: morphine, meth (methamphetamine), ketamine, cocaine, ecstasy (methylenedioxyamphetamine), marijuana (tetrahydrocannabinolic acid);
10. Have a history of any clinically serious disease or disease or condition that the investigator believes may affect the test results, including but not limited to a history of circulatory, endocrine, nervous system, digestive system, urinary system or blood, immune, psychiatric and metabolic diseases;
11. QTcF > 450 ms at screening or baseline 12-lead ECG (maximum retest 2 times allowed, average value can be taken), or there are other abnormalities judged by the investigator to be clinically significant;
12. Vital signs, physical examination, laboratory tests, abdominal ultrasound or chest imaging at screening, etc., suggest that there are abnormalities that are judged to be clinically significant by the investigator;
13. Within 4 weeks before randomization, positive hepatitis B surface antigen (HBsAg), or positive anti-hepatitis C virus (HCV) antibody, or positive human immunodeficiency virus (HIV) antibody, or positive syphilis antibody;
14. Use of any prescription drug, over-the-counter drug, Chinese herbal medicine or dietary supplement within 2 weeks prior to randomization;
15. Those who have participated in clinical trials of any other drug or medical device within 3 months before randomization or within 5 half-lives of the drug (subject to whether to administer or use the device);
16. Have received BCG vaccine within 12 months prior to screening; or vaccination or exposure to other live vaccines or live attenuated vaccines (except COVID vaccines) within 3 months prior to randomization; or those who plan to be vaccinated during the trial;
17. Those who have undergone any surgery within the 3 months prior to randomization, or who have not recovered after surgery, or who may have surgery or hospitalization plans during the estimated trial period;
18. Those who donate blood (or blood loss) within 3 months of randomization and donate blood (or blood loss) in an amount ≥ 400 mL, or receive blood transfusion;
19. The subject is judged by the investigator to have circumstances that affect the absorption, distribution, metabolism and excretion of the drug or can reduce compliance or other factors that are not suitable to participate in this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
SHR7280 and its main Pk parameter AUC0-t | Day 1 to Day 5
SHR7280 and its main Pk parameter AUC0-∞ | Day 1 to Day 5
SHR7280 and its main Pk parameter Cmax | Day 1 to Day 5
Relative bioavailability (F%) value between SHR7280 dry suspension and SHR7280 tablet: F% = AUC0-t (dry suspension) / AUC0-t (tablet) ×100% | Day 1 to Day 5

SECONDARY OUTCOMES:
SHR7280 and its main Pk parameter Tmax (SHR7280 only) | Day 1 to Day 5
SHR7280 and its main Pk parameter t1/2 (SHR7280 only) | Day 1 to Day 5
SHR7280 and its main Pk parameter CL/F (SHR7280 only) | Day 1 to Day 5
SHR7280 and its main Pk parameter Vz/F (SHR7280 only) | Day 1 to Day 5
Adverse events | Day 1 to Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu X, Qin R, Shu C, Shen K, Li X, Ma L, Li X, Li L, Peng J, Huang D, Chen S, Xie Z, Ye L, Duan L. Relative Bioavailability of Single-Dose Oral Administration of Two SHR7280 Formulations (Dry Suspension and Tablets) in Healthy Chinese Volunteers. Clin Drug Investig. 2025 Sep;45(9):643-650. doi: 10.1007/s40261-025-01470-7. Epub 2025 Aug 8. PMID 40779283